CLINICAL TRIAL: NCT04052256
Title: The Heartflow Coronary Disease Progression Evaluation Study
Acronym: THRONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Director of Interventional Cardiology, Erasmus Medical Center
Other Study IDs: THRONE1
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve; Coronary computed tomography angiography; Computational fluid dynamics; Plaque characteristics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intermediate coronary lesions: Patients (age ≥ 18 years) who have undergone invasive coronary angiography and have a minimum of one non-treated coronary artery with a measured invasive FFR of 0.81-0.90.
  Interventions: Diagnostic Test: Coronary computed tomography angiography

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography — Computational fluid dynamic model information derived from CT

SUMMARY:
Invasively measured fractional flow reserve (FFR) has proven to be useful in guiding coronary revascularization. Several studies have shown that it is justified to treat lesions with a value of 0.80 or lower and safe to defer from PCI in lesions with a value of >0.80. Recently, computational fluid dynamics have allowed FFR measurement from coronary computed tomography angiography images (FFRCT) with excellent diagnostic accuracy compared to invasive FFR.

FFRCT can also effectively guide revascularization safely deferring patient with FFRCT >0.80 from invasive angiography. In functionally non-significant lesions, computational fluid dynamic models in addition to CT plaque characteristics (low attenuation, positive remodelling, spotty calcification and napkin-ring sign) may be able to predict which lesions will become flow-limiting, causing clinical events in the future.

This study will evaluate disease progression in intermediate lesions (invasive FFR 0.81-0.90 at baseline) using FFRCT at 2 years and determine whether CT characteristics may help to identify lesions that are more susceptible for FFR decline. Additionally, we will correlate CT characteristics with coronary events (a composite endpoint consisting of all-cause mortality, target-vessel myocardial infarction and clinically driven target-vessel revascularization) up to 5 years after the baseline invasive FFR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (age ≥ 18 years) treated with PCI (for non-ST elevation myocardial infarction, unstable or stable angina and silent ischemia) or who undergo invasive FFR.
2. Minimum of one non-treated coronary artery with an intermediate lesion and invasive FFR 0.81-0.90 to serve as the target vessel for FFRCT.

Exclusion Criteria:

1. ST elevation myocardial infarction.
2. Previous CABG.
3. Target vessel for FFR measurement < 2.0 mm in diameter.
4. Contraindications to contrast agents, beta-blocking agents, nitroglycerin or adenosine.
5. Life expectancy less than 3 years.
6. Creatinine clearance < 30 ml/min*1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (age ≥ 18 years) treated with PCI (for non-ST elevation myocardial infarction, unstable or stable angina and silent ischemia) or who undergo invasive FFR.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Coronary atherosclerotic disease progression | 2 years
  FFRCT

SECONDARY OUTCOMES:
Target lesion failure Target vessel failure | 3-5 years
  Composite of all-cause mortality, target-vessel myocardial infarction and cinically driven target vessel revascularization.
Any coronary revascularisation | 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Leipsic, MD, PhD, Study Chair — University of British Columbia
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No